CLINICAL TRIAL: NCT01247584
Title: Telomere Length and Telomerase Mutations in Pediatric Acute Myeloid Leukemia
Brief Title: Biomarkers in Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B2; COG-AAML11B2 (Other: Children's Oncology Group); NCI-2011-02846 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies; childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute myeloblastic leukemia without maturation (M1); childhood acute myelomonocytic leukemia (M4); childhood acute myeloblastic leukemia with maturation (M2)
MeSH Terms: conditions — Leukemia | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying bone marrow samples from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the frequency of germline telomerase mutations in pediatric patients with acute myeloid leukemia (AML) demonstrating prolonged myelosuppression, defined as ≥ 1 episode > 35 days of neutrophil count recovery after chemotherapy, to the pediatric patients with the expected myelosuppression, defined as consistently < 35 days of neutrophil count recovery after chemotherapy.
* To assess association between telomerase mutations and incidence of grade 3 or 4 mucositis, relapse, and death.
* To compare germline (remission) telomere length in pediatric AML patients demonstrating delayed bone marrow recovery with the pediatric patients with consistently expected recovery.
* To assess whether a correlation between telomere length and incidence of grade 3 or 4 mucositis, relapse, and death exist.

OUTLINE: This is a multicenter study.

Cryopreserved bone marrow samples are analyzed for DNA sequencing and mutation by Sanger-based sequencing methods, quantitative PCR, and SeqMan Pro (Lasergene from DNAStar). Results are then compared with previously published data and existing databases to determine the allele frequency in control populations.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Enrolled on CCG-2961 and meeting 1 of the following criteria:

  * More than 35 days to recover to an ANC > 500/mm³ after any course of chemotherapy
  * Consistently recovered < 35 days to an ANC > 500/mm³ after all courses of chemotherapy
* Available cryopreserved cell from diagnostic and end-of-therapy samples

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of mutations
Relapse-free survival
Overall survival
Difference in telomere length

CONTACTS AND LOCATIONS:
Overall Officials: Maria M. Gramatges, MD, Principal Investigator — Baylor College of Medicine